CLINICAL TRIAL: NCT06963619
Title: NTproBNP2 Test Kit (Time-Resolved Immunofluorescence Method) Reference Interval Establishment Study Protocol
Brief Title: AQT90 FLEX NTproBNP (N-terminal Pro-brain Natriuretic Peptide) 2 Test Kit - Reference Interval Study Protocol - China
Status: Not yet recruiting | Type: Observational
Sponsor: Radiometer Medical ApS (Industry)
Responsible Party: Sponsor
Other Study IDs: DC-088045
Record Dates: First submitted 2025-04-21; First posted 2025-05-09 (Actual); Last update posted 2025-05-09 (Actual); Status verified 2025-01

CONDITIONS: Diagnostic Tests

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
To establish the reference range of the NTproBNP2 Test Kit (time-resolved immunofluorescence method) in apparently healthy Chinese population.

ELIGIBILITY:
Inclusion Criteria:

Subjects who meet all the following criteria are eligible for inclusion:

1. Voluntarily participate in this study and sign informed consent;
2. Body Mass Index (BMI) ≥18.5 and <28kg/ m2;
3. Age ≥18 years old;
4. Through the investigator's consultation with the subjects, evaluate the subjects who meet the requirements of the reference individual of this study (refer to the "reference individual questionnaire").

Exclusion Criteria:

Subjects who meet any of the following criteria will be excluded:

1. Physical examination, laboratory test/examination results meet any of the following:

   * eGFR(estimated glomerular filtration rate) (formula: CKD-EPI, chronic kidney disease epidemiology collaboration) < 60 mL/min/1.732
   * Systolic blood pressure ≥130 mm Hg and/or diastolic blood pressure ≥80 mmHg
   * Glycated hemoglobin A1c (HbA1c) ≥ 6.0%; or fasting blood glucose ≥ 7.0 mmol/L
   * Total cholesterol ≥ 6.22 mmol/L and/or triglycerides ≥ 2.26 mmol/L
   * High-sensitivity troponin: Female: ≥15.6 pg/mL (ng/L), Male: ≥34.2 pg/mL (ng/L)
   * Electrocardiogram, with obvious abnormalities such as those that may cause cardiac structural changes or risk factors for arrhythmia as assessed by the investigator
2. Subjects who are unable to provide a sufficient volume (≈2 mL) of EDTAanticoagulated whole blood sample;
3. Subjects who withdraw informed consent;
4. Subjects assessed by the investigator as unsuitable for inclusion in this study.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: To establish the reference range of the NTproBNP2 Test Kit (time-resolved immunofluorescence method) in apparently healthy Chinese population.
Sampling Method: Non-Probability Sample
Enrollment: 240 (Estimated)
Dates: Start 2025-05 (Estimated); Primary Completion 2025-08 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
AQT90 FLEX NTproBNP2 Test Kit - Reference Interval Establishment - China | 12 months
  To establish the reference range of the NTproBNP2 Test Kit (time-resolved immunofluorescence method) in apparently healthy Chinese population.